CLINICAL TRIAL: NCT06262113
Title: A Decentralized Clinical Trial to Promote Evidence-Based Care for Underserved Patients With Neurofibromatosis 1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Vanessa Merker, PhD, Assistant Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024P000392; AD-2022C2-24790 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Neurofibromatosis 1
Keywords: Neurofibromatosis; NF1; Guideline; Healthcare; PCP; Parent; Pediatric; Primary Care; Annual Care; Physical Exam; Well-Child
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibromatoses

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental)
  Interventions: Other: Letters about NF1 Care (Content Type 1)
- Enhanced Usual Care Arm (Experimental)
  Interventions: Other: Letters about NF1 Care (Content Type 2)

INTERVENTIONS:
Other: Letters about NF1 Care (Content Type 1) — Participants will receive two letters about NF1 care, one for themselves and one for their primary care clinician, to read in advance of the patient's annual wellness visit
  Arms: Intervention Arm
Other: Letters about NF1 Care (Content Type 2) — Participants will receive two letters about NF1 care, one for themselves and one for their primary care clinician, to read in advance of the patient's annual wellness visit
  Arms: Enhanced Usual Care Arm

SUMMARY:
The goal of this fully decentralized, randomized controlled trial is to compare the efficacy of two educational interventions for individuals with Neurofibromatosis 1 (NF1). The primary objective of the study is to determine which intervention leads to higher rates of evidenced-based health screenings for NF1 patients in primary care settings.

Adults with NF1 and parents/guardians of children with NF1 from across the U.S. who do not go to a specialized NF clinic and who have an upcoming annual wellness visits (e.g. an annual physical, a well-child visit, etc.) scheduled with a primary care provider (PCP) are eligible to enroll in the study. To see if you might be eligible, fill out a prescreening survey here: https://redcap.link/mynfguide

DETAILED DESCRIPTION:
Background: The majority of individuals with Neurofibromatosis 1 (NF1) in the United States lack access to specialized NF1 clinics and consequently don't receive care aligned with national recommendations. To address this gap in care, researchers are evaluating two interventions to determine which one helps people get recommended NF1-related health screenings at their annual wellness visit with a primary care provider.

Methods: Participants (adult patients or parents) who enroll in the study will complete baseline survey assessments online before their PCP visit and then be randomized to one of two groups. Both groups will be given letters, one for themselves and one for their clinician, that describe NF1 care recommendations. After attending their annual wellness visit, all participants will be asked to complete an online follow-up survey. A small subsample of participants will also be asked to do a virtual qualitative interview. No visits to Massachusetts General Hospital are required for this study.

ELIGIBILITY:
Adult Inclusion Criteria:

* Currently lives in the United States (including Puerto Rico and other United States territories)
* Has a clinical diagnosis of neurofibromatosis 1
* Does not attend an NF clinic within the Children's Tumor Foundation NF Clinic Network
* Has an in-person, well-person visit with a primary care provider scheduled within 3 months of their consent
* Speaks English or Spanish

Parent/Guardian of a Child with NF1 Inclusion Criteria:

* Currently lives in the United States (including Puerto Rico and other United States territories)
* Cares for a child (age <18 years) with a clinical diagnosis of neurofibromatosis 1
* Does not attend an NF clinic within the Children's Tumor Foundation NF Clinic Network
* Their child has an in-person, well-person visit with a primary care provider scheduled within 3 months of their consent
* Speaks English or Spanish

Exclusion Criteria:

* Only one person per household may participate in the study
* Unwilling or unable to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Receipt of Recommended NF1 Health Screenings | 2 weeks after PCP visit
  Number of AAP and ACMG recommended health screenings received by the person with NF1 at the annual wellness visit with their PCP, as assessed by patient/parent self-report

SECONDARY OUTCOMES:
Patient Activation Measure® | At baseline and 2 weeks after PCP visit
  The Patient Activation Measure will be used to assess patient's and parent's self-efficacy managing their or their child's care. The patient form has 13 items and the parent form has 10 items. The measure has scores ranging from 0-100, where higher scores indicate higher patient/parent activation (e.g. self-efficacy in managing your own or your child's healthcare).
Consumer Assessment of Healthcare Providers and Systems (CAHPS®) Clinician and Group Survey Version 4.0 (Beta): Rating of the Visit | 2 weeks after PCP visit
  The CAHPS® Rating of the Visit will be used to assess patient/parent satisfaction with the visit. This rating is a single item scored from 0 to 10, where higher scores indicated a better visit.
Consumer Assessment of Healthcare Providers and Systems (CAHPS®) Clinician and Group Survey Version 4.0 (Beta): How Well Providers Communicate With Patients Subscale | 2 weeks after PCP visit
  The subscale will be used to assess How Well Providers Communicate With Patients. This scale will be scored from 0 to 100, where higher scores indicated better communication with patients.
Consumer Assessment of Healthcare Providers and Systems (CAHPS®) Clinician and Group Survey Version 4.0 (Beta): Providers' Use of Information to Coordinate Patient Care Subscale | 2 weeks after PCP visit
  The subscale will be used to assess Providers' Use of Information to Coordinate Patient Care. This scale will be scored from 0 to 100, where higher scores indicate better use of information to coordinate care.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Merker, PhD, Principal Investigator — Massachusetts General Hospital; Scott Plotkin, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to submit their complete de-identified data set to the Patient-Centered Outcomes Data Repository (PCODR) at the Inter-university Consortium for Political and Social Research (ICPSR) per PCORI guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The PCORI-designated repository will make the data available for third-party requests when PCORI makes the Final Research Report available on the PCORI website pursuant to PCORI's Process for Peer Review of Primary Research and Public Release of Research Findings, or at the time of publication of the research project's primary results in a peer-reviewed journal, whichever comes first.
Access Criteria: Individual investigators or teams of investigators seeking access to data from PCORI-funded studies must complete and submit a data request form to the PCORI-designated repository.
URL: https://www.pcori.org/about/governance/pcoris-policy-data-management-and-data-sharing

REFERENCES:
- [Background] Merker VL, Ma Y, Chibnik LB, Radtke HB, Kelts K, Yohay K, Ullrich NJ, Plotkin SR, Jordan JT. Self-reported access to specialty clinics and receipt of health surveillance among U.S. patients with neurofibromatosis 1: a national survey. Orphanet J Rare Dis. 2025 Apr 16;20(1):185. doi: 10.1186/s13023-025-03677-5. PMID 40241092
- [Background] Merker VL, Dai A, Radtke HB, Knight P, Jordan JT, Plotkin SR. Increasing access to specialty care for rare diseases: a case study using a foundation sponsored clinic network for patients with neurofibromatosis 1, neurofibromatosis 2, and schwannomatosis. BMC Health Serv Res. 2018 Aug 29;18(1):668. doi: 10.1186/s12913-018-3471-5. PMID 30157837
- [Background] Merker VL, Knight P, Radtke HB, Yohay K, Ullrich NJ, Plotkin SR, Jordan JT. Awareness and agreement with neurofibromatosis care guidelines among U.S. neurofibromatosis specialists. Orphanet J Rare Dis. 2022 Feb 10;17(1):44. doi: 10.1186/s13023-022-02196-x. PMID 35144646